CLINICAL TRIAL: NCT01961674
Title: Infrared Thermal Imaging for Assessing the Effect of Capsinoids on Brown Adipose Tissue Activity.
Brief Title: Studying the Effect of Capsinoids on Brown Fat Using Infrared Thermal Imaging.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Principal Investigator, Melvin Leow, Associate Professor, Singapore Institute of Food and Biotechnology Innovation
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 2013/00785
Record Dates: First submitted 2013-10-10; First posted 2013-10-11 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-02

CONDITIONS: Obesity; Diabetes; Impaired Glucose Tolerance
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Glucose Intolerance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Capsinoid arm (Experimental): On capsinoids
  Interventions: Dietary Supplement: Capsinoid/placebo and rice
- Placebo arm (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Capsinoid/placebo and rice

INTERVENTIONS:
Dietary Supplement: Capsinoid/placebo and rice — The subject will ingest six capsinoid/placebo capsules and a standardized amount of white rice (equivalent to 50g carbohydrates). Each capsule consists 1.5mg of capsinoids, making a total dose of 9mg capsinoids.

SUMMARY:
The primary hypothesis of this study is that consumption of capsinoids increases brown adipose tissue activity, detectable by infrared thermal imaging.

The secondary hypothesis is that consumption of capsinoids can affect an individual's glycaemic response.

DETAILED DESCRIPTION:
It has been recently established that brown adipose tissue (BAT) exists in adult humans. BAT is a thermogenic tissue which dissipates energy as heat. The primary objective of this study is to use thermal imaging to assess the effect of capsinoids on BAT activity in adult humans, and whether there is a relationship between the increase in energy expenditure and BAT activity after capsinoids intake. The secondary objective is to investigate whether capsinoids will have an effect on an individual's glycaemic response. Lean, healthy male volunteers will be recruited. There will be two test sessions which are randomized, where subjects will consume either capsinoids or placebo capsules, and a standardized amount of white rice (equivalent to 50g carbohydrates). Indirect calorimetry will be used to assess energy expenditure before and after consumption of the test meal. Thermal imaging of supraclavicular BAT, the primary BAT depot in humans, will be undertaken using an infrared thermal camera to assess changes in BAT temperature. Blood glucose levels will be monitored by finger prick blood sampling method. This study aims to investigate whether capsinoids consumption leads to changes in BAT temperatures detectable by the infrared thermal camera, to confirm the feasibility of using thermal imaging as a rapid, noninvasive, and reproducible way of studying BAT activity thus providing a platform to advance research in this emerging field of human BAT.

ELIGIBILITY:
Inclusion Criteria:

* Chinese ethnicity
* Male
* Healthy
* Age 21 - 30 years
* BMI 18.0 - 22.9 kg/m2
* Not on any prescribed medication
* Infrequent spicy food or chilli user (less than 3 times per week)

Exclusion Criteria:

* Smoker
* Fasting blood glucose > 5.5 mmol/L
* Resting blood pressure > 140/90 mmHg
* Any major medical conditions including diabetes, hypertension, cardiovascular disease, thyroid disorders
* Allergic or intolerant to foods presented in the study

Ages: 21 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Temperature at supraclavicular region | 2.5 hours post-consumption
  The temperature at the supraclavicular region following consumption of capsinoids will be determined using infrared thermal imaging.

SECONDARY OUTCOMES:
Glycaemic response | 2.5 hours post-consumption
  The blood glucose response to capsinoids measured over 2.5 hours following their consumption.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Nutrition Research Centre, Singapore, Singapore